CLINICAL TRIAL: NCT05756257
Title: Blood Pressure Variability and Ischemic Stroke Outcome
Acronym: BP-VISO
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: University of Chicago (Other); Massachusetts General Hospital (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00065750; 2000034922 (Other: Yale IRB); 1R01NS130189-01 (NIH)
Record Dates: First submitted 2023-02-15; First posted 2023-03-06 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Acute Ischemic Stroke; Blood Pressure Variability
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Ischemic Stroke: Blood pressure variability will be measured in the patients with acute ischemic stroke.

SUMMARY:
The goal of this observational study is to evaluate the role of blood pressure (BPV) variability in patients suffering from acute ischemic stroke. The main questions it aims to answer are:

1. To determine the association of BPV with functional/cognitive outcome after ischemic stroke.
2. To determine a pathophysiologic mechanism of BPV's deleterious effect on functional outcome.
3. To evaluate potential treatment targets to pharmacologically reduce BPV after ischemic stroke.

DETAILED DESCRIPTION:
Increased blood pressure variability (BPV) has consistently been associated with two to three times higher risk of disability or mortality after acute ischemic stroke (AIS) in retrospective analyses, independent of mean blood pressure. The investigators' central hypothesis is that increased BPV is harmful after AIS and warrants reduction. However, prior BPV research in AIS patients has been retrospective and limited by non-standardized BP measurement and, therefore, BPV is not mentioned in current stroke guidelines. To address the limitations of prior BPV research, determine mechanisms of BPV's deleterious effect, and identify potentially effective methods to reduce BPV, the proposed study will: 1) prospectively validate that "short-term" and "long-term" BPV after AIS onset is associated with functional outcome and define the effect size of different levels of BPV, 2) utilize portable MRI to confirm that final infarct volume is mechanistically related to BPV, and 3) utilize bedside pupillometry to determine how the autonomic nervous system contributes to BPV after AIS and evaluate the class effect of antihypertensive medications on BPV. To achieve these goals, the study will enroll 150 patients who have anterior circulation stroke and a baseline NIH Stroke Scale ≥4 within 48 hours of AIS onset at three study sites. With completion of the Aims, the study will define the outcome for a future trial, the effect size of BPV on individual outcomes and composites, the duration for lowering BPV (24-72 hours vs. weeks or months), and potential interventions to reduce BPV. Pharmacologic BPV reduction would be an inexpensive and widely available intervention, able to be administered in a range of healthcare settings. By completing the proposed aims, the investigators will be ideally positioned to test accessible targeted interventions to diminish the morbidity and mortality of AIS.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke according to the American Heart Association (AHA) definition and either:

  1. CT or MRI showing ischemic stroke in the anterior circulation (frontal, parietal or superior temporal lobes), or
  2. Occlusion of the internal carotid, middle cerebral or anterior cerebral arteries on computed tomography angiography (CTA) or magnetic resonance angiography (MRA)

     Onset of ischemic stroke within 48 hours and able to get baseline pMRI within 72 hours of arrival

     4) NIH Stroke Scale ≥ 4 at time of enrollment

     Exclusion Criteria:
* Pre-morbid mRS ≥3
* Predicted hospital system admission <72 hours
* Pacemaker or other MRI contraindications per American College of Radiology guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke serve as the source population for the study and will be identified as inpatients at participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in Functional outcome | 90 days and 1 Year
  Modified Rankin Scale, the scale uses a range of 0-6 where higher scores indicate decreased function.
Imaging outcome | 72 hours +/- 60 hours
  Final infarct volume on MRI at 72 hours

SECONDARY OUTCOMES:
Incidence of stroke | 90 days
  Incidence of new (recurrent) ischemic stroke
Incidence of stroke | 1 year
  Incidence of new (recurrent) ischemic stroke
Change in Montreal Cognitive Assessment scale (MoCA-BLIND) to assess post-stroke cognition | 3 days and 1 year
  Post-stroke cognition will be assessed using the MoCA-BLIND, The MoCA-BLIND assess six different cognitive domains (excludes visual stimulus) over the phone: memory, attention, language, abstraction, delayed recall, and orientation. The MoCA-BLIND is scored from 0-22. Lower scores indicate less cognitive impairment.
Change in Oral Trails A and B Test to assess post-stroke cognition | 3 days and 1 year
  Post-stroke cognition will be assessed using the Oral Trails A and B Test to measure psychomotor speed, visual search, and attention. The test is scored based on how many seconds it takes to complete each part. Higher scores indicate a higher degree of cognitive impairment.
Change in Category Fluency tests to assess post-stroke cognition | 3 days and 1 year
  Categorical verbal fluency tests (CFT) are used to assess the integrity of semantic memory in individuals with brain damage. Participants are given 1 min to produce as many unique words as possible within a semantic category (category fluency) or starting with a given letter (letter fluency). The participant's score in each task is the number of unique correct words.
Change in Patient Health Questionnaire (PHQ-9) to assess mood | 3 days and 1 year
  Nine items asking about the frequency of specific depressive symptoms experienced. The response options are scored from 0 to 3, indicating "not at all" to "nearly every day." The total score on the PHQ-9 ranges from 0 to 27, with higher scores indicating greater severity of depressive symptoms. The scoring can also be divided into categories, with scores of 0-4 indicating minimal or no depression, 5-9 indicating mild depression, 10-14 indicating moderate depression, 15-19 indicating moderately severe depression, and 20-27 indicating severe depression.
Change in General Anxiety Disorder-7 (GAD-7) to assess mood | 3 days and 1 year
  General Anxiety Disorder- 7 (GAD-7) is a 7 item self report instrument that measures anxiety Items are scored on a 4-point scale, ranging from "not at all (0)" to "nearly everyday (3)". Item scores are summed with a total score ranging from 0 to 21: 0-4 Minimal anxiety; 5-9 Mild anxiety; 10-14 Moderate anxiety; 15-21 Severe anxiety.
Change in Lawton Instrumental Activities of Daily Living (IADL) Scale to assess adaptive functioning | 3 days and 1 year
  The IADL assesses a person's ability to perform tasks such as using a telephone, doing laundry, and handling finances. It consists of 8 items and total score is achieve by summing all items. Each item is scored 0 = less able or 1 = more able. Total score range is from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men to avoid potential gender bias. The higher the score, the greater the person's abilities.
Change in Katz Index of Independence in Activities of Daily Living (ADL) to assess adaptive functioning | 3 days and 1 year
  The Katz IADL assesses the patient's need for assistance in performing basic activities of daily living. Total scores range from 0-12, with higher scores indicating better levels of functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Adam de Havenon, MD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No